CLINICAL TRIAL: NCT04204148
Title: Multivariate Analysis of Cough After Uniport Video-assisted Thoracoscopic Surgery Pneumonectomy
Brief Title: To Explore the Related Factors of Cough After Thoracoscopic Pneumonectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019113
Record Dates: First submitted 2019-12-14; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Cough
Keywords: postoperative cough; Multivariate analysis; non-small cell lung cancer (NSCLC); Uniport Video-assisted Thoracoscopic Surgery
MeSH Terms: conditions — Cough; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical characteristics of the patients: including sex,age,smoking history,tumor location and tumor diameter
- Logistic regression analysis of influencing factors of c: The Leicester Cough Questionnaire in Mandarin Chinese (LCQ-MC) was used to evaluate the degree of cough in patients. The LCQ-MC is divided into three dimensions: physical, psychological and social. There are a total of 19 questions, and each question has seven options (positive scoring, grades 1-7; the higher the score is, the lighter the cough).

SUMMARY:
To explore the related factors of cough after Uniport video-assisted thoracoscopic surgery pneumonectomy, and to provide theoretical basis and social accumulation of new knowledge for the diagnosis and treatment of cough after pneumonectomy in the future.

DETAILED DESCRIPTION:
Intractable cough after thoracoscopic pneumonectomy is one of the common complications after pneumonectomy. The incidence of cough can reach 25% ≤ 50%. Cough after operation can aggravate the pain of incision, prolong the hospitalization time, increase the cost of hospitalization, affect the conversation and even sleep of the patients, increase the psychological burden of the patients, and reduce the quality of life of the patients accordingly. Therefore, through this study, the investigators hope to understand the related factors of cough after thoracoscopic pneumonectomy and whether there are predictable risk factors, so as to provide theoretical basis for reducing the occurrence of cough after pneumonectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, male and female
* Uniport video-assisted thoracoscopic surgery
* No cough symptoms within two weeks before operation
* Informed consent form was signed before operation

Exclusion Criteria:

* Diabetes , heart, brain, liver and kidney diseases
* Chest radiographs / CT in recent months indicate pneumonia
* Pulmonary function cannot tolerate lobectomy / segmental / cuneiform resection
* Distant metastasis patients
* Before operation, there were internal causes of cough (including respiratory tract infectious diseases, pharyngitis, allergic rhinitis, posterior nasal drip syndrome, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years old, male and female
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The mean Leicester Cough Questionnaire in Mandarin Chinese (LCQ-MC) score before and after surgery | The day before surgery,two weeks after surgery,one month after surgery
  The Leicester Cough Questionnaire in Mandarin Chinese (LCQ-MC), which assesses the cough-related quality of life, consists of 19 items divided into three domains: the physical (8 items), psychological (7 items) and social (4 items) domains. A 7-point Likert scale was used to score individual domains. The total scores ranged from 3 to 21, with a higher score indicative of a better health status

SECONDARY OUTCOMES:
Hospitalization days | From the first days after surgery to discharge,up to 4 weeks
  The numbers of days of patients stay in the hospital after surgery
Drainage | Measure the volume every 24 hours,up to 4 weeks
  The total volume of fluid
Anesthesia time | Record total anesthesia during surgery
  Time from patient anesthesia to extubation

CONTACTS AND LOCATIONS:
Overall Officials: Liping Peng, Principal Investigator — The First Affiliated Hospital of Soochow University; Liuying Pan, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dicpinigaitis PV, Rauf K. The influence of gender on cough reflex sensitivity. Chest. 1998 May;113(5):1319-21. doi: 10.1378/chest.113.5.1319. PMID 9596313
- [Result] Birring SS, Spinou A. How best to measure cough clinically. Curr Opin Pharmacol. 2015 Jun;22:37-40. doi: 10.1016/j.coph.2015.03.003. Epub 2015 Mar 25. PMID 25819594
- [Result] Harle ASM, Blackhall FH, Molassiotis A, Yorke J, Dockry R, Holt KJ, Yuill D, Baker K, Smith JA. Cough in Patients With Lung Cancer: A Longitudinal Observational Study of Characterization and Clinical Associations. Chest. 2019 Jan;155(1):103-113. doi: 10.1016/j.chest.2018.10.003. Epub 2018 Oct 13. PMID 30321508
- [Result] Brignall K, Jayaraman B, Birring SS. Quality of life and psychosocial aspects of cough. Lung. 2008;186 Suppl 1:S55-8. doi: 10.1007/s00408-007-9034-x. Epub 2007 Oct 16. PMID 17939003
- [Result] Xie MR, Zhu YF, Zhou MQ, Wu SB, Xu GW, Xu SB, Xu MQ. Analysis of factors related to chronic cough after lung cancer surgery. Thorac Cancer. 2019 Apr;10(4):898-903. doi: 10.1111/1759-7714.13021. Epub 2019 Mar 15. PMID 30875149
- [Result] Koskela HO, Latti AM, Pekkanen J. The impacts of cough: a cross-sectional study in a Finnish adult employee population. ERJ Open Res. 2018 Nov 12;4(4):00113-2018. doi: 10.1183/23120541.00113-2018. eCollection 2018 Oct. PMID 30443552
- [Result] Wang P, Zhu M, Zhang D, Guo XG, Zhao S, Zhang XL, Wang DL, Liu CT. The relationship between chronic obstructive pulmonary disease and non-small cell lung cancer in the elderly. Cancer Med. 2019 Aug;8(9):4124-4134. doi: 10.1002/cam4.2333. Epub 2019 Jun 11. PMID 31184445
- [Derived] Pan LY, Peng LP, Xu C, Ding C, Chen J, Wang WY, Zhu XY, Zhao J, Li C. Predictive factors of cough after uniportal video-assisted thoracoscopic pulmonary resection. J Thorac Dis. 2020 Oct;12(10):5958-5969. doi: 10.21037/jtd-20-2652. PMID 33209428